CLINICAL TRIAL: NCT04464629
Title: Assessing the Efficacy and Safety of DEXTENZA, Sustained Release Dexamethasone 0.4 mg Insert, When Placed Within the Lower Eye Lid Canaliculus in Pseudo Phakic Patients Undergoing Gas Bubble Repair and Laser Following Retinal Detachment
Brief Title: Assessing the Efficacy and Safety of DEXTENZA in Pseudo Phakic Patients Undergoing Gas Bubble Repair and Laser Following Retinal Detachment
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Midwest Eye Institute (Other)
Collaborators: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Principal Investigator, Neil Finnen, MD, Principal Investigator, Midwest Eye Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: The FINNEN Study
Record Dates: First submitted 2020-07-06; First posted 2020-07-09 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Retinal Detachment
MeSH Terms: conditions — Retinal Detachment | interventions — Calcium Dobesilate; prednisolone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intracanalicular Sustained Release Dexamethasone, 0.4 mg (Experimental): Intracanalicular dexamethasone insert contains 0.4 mg dexamethasone and is designed to provide a sustained and tapered release of therapeutic levels of dexamethasone to the ocular surface for up to 30 days for the reduction of post-surgical inflammation and pain associated with ocular surgery.
  Interventions: Drug: Dextenza
- topical prednisolone acetate 1%. (Active Comparator)
  Interventions: Drug: Prednisolone Acetate

INTERVENTIONS:
Drug: Dextenza — Intracanalicular sustained release dexamethasone insert 0.4 mg
  Arms: Intracanalicular Sustained Release Dexamethasone, 0.4 mg
Drug: Prednisolone Acetate — Topical Prednisolone acetate 1% ophthalmic suspension
  Arms: topical prednisolone acetate 1%.

SUMMARY:
This prospective, open-label, single-center, randomized, investigator-sponsored clinical study seeks to investigate: how will pseudophakic patients respond in terms of objective and subjective outcomes, when treated with Dextenza compared to topical prednisolone acetate following gas bubble repair and laser for RD.

DETAILED DESCRIPTION:
Subjects who have given informed consent and determined to be eligible at screening will be randomized in a 1:1 ratio to DEXTENZA (placed once in the lower punctum) or the use of topical Prednisolone acetate 1% drops (four times daily). They will be observed for a period of 3-months for both pain and inflammation of the eye.

ELIGIBILITY:
Inclusion Criteria:

* Pseudophakic
* Retinal Detachment
* Age 18 years and older
* Scheduled for gas bubble repair and laser surgery following retinal detachment
* Willing and able to comply with clinic visits and study related procedures
* Willing and able to sign the informed consent form

Exclusion Criteria:

* Patients under the age of 18.
* Pregnancy (must be ruled out in women of child-bearing age with pregnancy test)
* Active infectious systemic disease
* Active infectious ocular or extraocular disease
* Obstructed nasolacrimal duct in the study eye(s)
* Hypersensitivity to dexamethasone
* Patients being treated with immunomodulating agents in the study eye(s)
* Patients being treated with immunosuppressants and/or oral steroids
* Patients with severe disease that warrants critical attention, deemed unsafe for the study by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Mean change in pain score | 30 Days
  Average change in pain based on whats reported on the Ocular Pain Assessment
Post-op pain scores | 30 Days
  Ocular Pain Assessment: Measured on a scale from 0-10 where 0 (minimum) is no pain and 10 (maximum) is extreme pain. High reported pain means a worse outcome.

SECONDARY OUTCOMES:
Mean change in anterior chamber cell and flare score | 30 days
  Post op inflammation scores as measured on a scale of 0-4: Anterior Chamber Cell Count (Absence of cell to be defined as a grade of: 0-0.5, 4 being the maximum) and Anterior Chamber Flare Score (0 is the minimum, and 4 is the maximum). High reported cell and flare means a worse outcome.
Cystoid Macular Edema | 30 days
  Amount of central thickness macular swelling as measured by Optical Coherence Tomography (OCT)
Best Corrected Visual Acuity | 90 days
  As measured on ETDRS
Physician Ease of Dextenza insertion | Day 1
  The investigator will grade the level of ease of insertion of the intracanalicular insert on a 0 to 10-point (0 being the minimum and 10 being the maximum) scale with 0 being very easy insertion and 10 being very hard. Difficult insertion means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Finnen, MD, Principal Investigator — Midwest Medical Advisors, Inc
Locations (1):
- Midwest Eye Institute, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No